CLINICAL TRIAL: NCT00187954
Title: Retinal Photography in Women With Chest Pain: A WISE/ARIC Collaboration
Brief Title: WISE ARIC: Retinal Photography in Women With Chest Pain
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: WISE ARIC; HL64924
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Chest Pain
Keywords: women; chest pain; microvascular dysfunction; retinal photography; Retinal vascular function
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purposes of this study are:

* To correlate the severity of retinal arteriolar narrowing and other microvascular changes, as determined from retinal photographs and video imaging, to measures of coronary microvascular function in women evaluated for chest pain.
* To evaluate measures of vascular compliance with applanation tonometry and photoplethysmography using a nasal alar probe.

DETAILED DESCRIPTION:
Women who meet study eligibility criteria and provide written informed consent will have a baseline physical exam, including measurements of heart rate, blood pressure, weight. Medical history will be updated, specifically cardiovascular events (hospitalizations, procedures) since last contact and current medications. Patients will be scheduled for retinal photography. Those who are currently being screened and qualify for EWISE or other ancillary studies will have retinal photography scheduled as close to the index CFR as possible and prior to receiving randomized therapy.

The retinal photography will follow a standardized written protocol.

For the second protocol, 100 patients will be scheduled for an appointment in the Eye clinic where they will meet the Women's Ischemic Syndrome Evaluation (WISE)/Atherosclerosis Risk in Communities (ARIC) staff and complete the baseline information and have a brief physical examination. They will then have provocative testing completed with retinal imaging.

ELIGIBILITY:
Inclusion Criteria:

* Women who participated in or are being screened for the WISE or EWISE or any ancillary studies
* Willing to provide written informed consent
* Have recorded measurements of coronary flow reserve, with or without obstructive coronary disease

Exclusion Criteria:

* Unwilling to complete study required procedures
* Contraindication to adenosine

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who participated in or are being screened for the WISE or EWISE or any ancillary studies
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2003-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Arteriole to venule ratio (AVR) | baseline
  retinal arteriolar and venule diameters reflected as a ratio

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Handberg, PHD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Wattanakit K, Folsom AR, Chambless LE, Nieto FJ. Risk factors for cardiovascular event recurrence in the Atherosclerosis Risk in Communities (ARIC) study. Am Heart J. 2005 Apr;149(4):606-12. doi: 10.1016/j.ahj.2004.07.019. PMID 15990741